CLINICAL TRIAL: NCT07099820
Title: Role of Indexed Oxygen Delivery in Anastomotic Insufficiencies in Elective Laparoscopic Colorectal Resections for Cancer: a Prospective Observational Cohort Study
Brief Title: Role of Indexed Oxygen Delivery in Anastomotic Insufficiencies in Elective Laparoscopic Colorectal Resections for Cancer
Status: Recruiting | Type: Observational
Sponsor: Saint Camillus International University of Health Sciences (Other)
Responsible Party: Principal Investigator, Diego Fiume, Principal Investigator, Saint Camillus International University of Health Sciences
Other Study IDs: 00154/20
Record Dates: First submitted 2025-07-22; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anastomosis; Complications; Anastomosis, Surgical; Anastomosis, Leaking; Anastomotic Leaks; Anastomotic Failure of Flap; Anastomotic Leak Large Intestine; Anastomotic Complication; Anastomotic Dehiscence in Colorectal Surgery; Anastomotic Leakage in Colon Surgery; Oxygen Delivery; Oxygen Delivery (DO2)
Keywords: anastomosis; anastomotic leaks; anastomosis leaking; colorectal surgery; colon surgery; oxygen delivery; DO2; DO2I; non-invasive monitoring
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from neoplasm of the colo-rectum: Patients underwent colic resection

SUMMARY:
Colorectal cancer is a very commonly diagnosed malignancy worldwide, and surgical resection remains the mainstay of treatment. Outcomes depend on preoperative staging, surgical quality, complication rates, and multidisciplinary care; minimally invasive techniques have reduced local and systemic complications. However, anastomotic dehiscence (AD) remains the most significant local complication.

AD is a breach in the anastomotic integrity creating a communication between intra- and extra-luminal compartments. Mortality rates vary from 1.7% to 29%.

Reduced oxygen delivery-pre-, intra-, or post-operatively-can contribute to AD, while adequate oxygenation improves healing. Supplemental O₂ (FiO₂ 80%) has been shown to reduce AD risk after gastric surgery.

Tissue oxygen delivery can be quantified by indexed oxygen delivery (DO2I), defined as ml/min/m² and determined by cardiac output, hemoglobin, and saturation. Pulse cardiac output (CO)-Oximeter® (Masimo), allow continuous non-invasive monitoring of these parameters.

This prospective observational cohort study aims to explore the correlation between intraoperative DO2I and the risk of postoperative anastomotic dehiscence, using the non-invasive technologies described.

DETAILED DESCRIPTION:
Colorectal cancer is the third most commonly diagnosed malignancy worldwide, accounting for ~10% of all cancers and ranking as the fourth leading cause of cancer death, with 1.9 million new cases and ~930,000 deaths in 2020. Surgical resection remains the mainstay of treatment for nonmetastatic cases and plays a crucial role in managing metastatic disease. Outcomes depend on preoperative staging, surgical quality, complication rates, and multidisciplinary care. Since Jacobs' 1991 report of 20 laparoscopic resections, minimally invasive techniques have reduced local and systemic complications. However, anastomotic dehiscence (AD) remains the most significant local complication, increasing hospital stays, costs, morbidity, mortality, and negatively affecting overall prognosis.

The International Study Group of Rectal Cancer defines AD as a breach in the anastomotic integrity creating a communication between intra- and extra-luminal compartments. Mortality rates vary widely, from 1.7% in an Australian cohort to as high as 29% in other reports, with AD accounting for roughly one-third of postoperative colorectal surgery deaths. Incidence is site-dependent: 1-20% in colo-rectal, 0-2% in colo-colic, and 0.02-4% in ileo-colic anastomoses.

Risk factors are categorized as local or systemic. Local factors include anastomotic level, technique (mechanical vs. manual), surgeon experience, bowel prep, use of laparoscopy, diverting stomas, drains, radiotherapy, chemotherapy, and gut microbiota. Systemic factors include male sex, malnutrition, hypoalbuminemia, anemia, comorbidities, American Society of Anesthesiologists (ASA) score, nonsteroidal anti-inflammatory drug (NSAID) use, smoking, alcohol, peripheral vascular disease, obesity, and diabetes. Reduced oxygen delivery-pre-, intra-, or post-operatively-can contribute to AD, while adequate oxygenation improves healing. Supplemental O₂ (FiO₂ 80%) has been shown to reduce AD risk after gastric surgery.

Tissue oxygen delivery can be quantified by indexed oxygen delivery (DO2I), defined as ml/min/m² and determined by cardiac output, hemoglobin, and saturation. A DO2I < 400 ml/min/m² is associated with increased AD risk; normal values range from 450-550 ml/min/m². Below this, compensation through increased extraction fails beyond a critical threshold, leading to anaerobic metabolism and lactic acidosis. Accurate DO2I calculation requires cardiac output monitoring.

While the esophageal Doppler is the standard for cardiac output measurement, its invasiveness and operator dependence limit use. Less invasive alternatives, like pulse-contouring (e.g., PiCCO, Vigileo) or fully non-invasive methods like ClearSight®, offer continuous hemodynamic data. ClearSight® uses the volume-clamp method via a finger cuff and photoplethysmography to measure real-time arterial pressure and advanced parameters such as cardiac output and stroke volume.

DO2I calculation also requires hemoglobin levels, which fluctuate intraoperatively due to blood loss and fluid shifts. Reliable measurement would ideally involve repeated blood sampling, which adds invasiveness and cost. Advances in pulse oximetry, like the Rad-97 Pulse CO-Oximeter® (Masimo), allow continuous non-invasive monitoring of O₂ saturation, Hb, carboxyhemoglobin, methemoglobin, perfusion index, and more, even under low perfusion or motion conditions.

This prospective observational cohort study aims to explore the correlation between intraoperative DO2I and the risk of postoperative anastomotic dehiscence, using the non-invasive technologies described.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * Candidates for elective laparoscopic colo-rectal surgery for neoplastic pathology with ileo-colic, colo-colic and colo-rectal anastomosis.

Exclusion Criteria:

* • Age < 18 years

  * Inability to give valid informed consent
  * Candidates for operations involving other wards
  * Candidates for emergency surgery
  * Candidates for laparotomic surgery
  * Colo- or ileo-stomy
  * Contraindications to the use of the volume clamp system for haemodynamic monitoring (conditions with significant alteration of finger perfusion, such as Raynaud's disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Generale Surgery, St.Eugenio Hospital, Rome, Italy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative anastomotic dehiscence | perioperatively
  Breach in the anastomotic integrity creating a communication between intra- and extra-luminal compartments

SECONDARY OUTCOMES:
Length of Stay | perioperatively
  Days in hospital
Transfusions | perioperatively
  Number of blood units transfused
Mortality | perioperatively
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Diego Fiume, MD PhD, Study Chair — UniCamillus - Saint Camillus International University of Health and Medical Sciences
Locations (1):
- St. Eugenio Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant Data (IPD); however, anonymized data may be made available upon reasonable request, subject to sponsor approval and ethical considerations.

REFERENCES:
- [Background] Sciuto A, Merola G, De Palma GD, Sodo M, Pirozzi F, Bracale UM, Bracale U. Predictive factors for anastomotic leakage after laparoscopic colorectal surgery. World J Gastroenterol. 2018 Jun 7;24(21):2247-2260. doi: 10.3748/wjg.v24.i21.2247. PMID 29881234
- [Background] Krarup PM, Nordholm-Carstensen A, Jorgensen LN, Harling H. Anastomotic leak increases distant recurrence and long-term mortality after curative resection for colonic cancer: a nationwide cohort study. Ann Surg. 2014 May;259(5):930-8. doi: 10.1097/SLA.0b013e3182a6f2fc. PMID 24045445
- [Background] Alvandipour M, Mokhtari-Esbuie F, Baradari AG, Firouzian A, Rezaie M. Effect of Hyperoxygenation During Surgery on Surgical Site Infection in Colorectal Surgery. Ann Coloproctol. 2019 Feb;35(1):9-14. doi: 10.3393/ac.2018.01.16. Epub 2019 Feb 28. PMID 30879279
- [Background] Shoemaker WC, Appel PL, Kram HB, Waxman K, Lee TS. Prospective trial of supranormal values of survivors as therapeutic goals in high-risk surgical patients. Chest. 1988 Dec;94(6):1176-86. doi: 10.1378/chest.94.6.1176. PMID 3191758
- [Background] Levy BF, Fawcett WJ, Scott MJ, Rockall TA. Intra-operative oxygen delivery in infusion volume-optimized patients undergoing laparoscopic colorectal surgery within an enhanced recovery programme: the effect of different analgesic modalities. Colorectal Dis. 2012 Jul;14(7):887-92. doi: 10.1111/j.1463-1318.2011.02805.x. PMID 21895923
- [Background] Sangkum L, Liu GL, Yu L, Yan H, Kaye AD, Liu H. Minimally invasive or noninvasive cardiac output measurement: an update. J Anesth. 2016 Jun;30(3):461-80. doi: 10.1007/s00540-016-2154-9. Epub 2016 Mar 9. PMID 26961819
- [Background] Ameloot K, Palmers PJ, Malbrain ML. The accuracy of noninvasive cardiac output and pressure measurements with finger cuff: a concise review. Curr Opin Crit Care. 2015 Jun;21(3):232-9. doi: 10.1097/MCC.0000000000000198. PMID 25922896
- [Background] Schietroma M, Cecilia EM, Carlei F, Sista F, De Santis G, Piccione F, Amicucci G. Prevention of anastomotic leakage after total gastrectomy with perioperative supplemental oxygen administration: a prospective randomized, double-blind, controlled, single-center trial. Ann Surg Oncol. 2013 May;20(5):1584-90. doi: 10.1245/s10434-012-2714-7. Epub 2012 Oct 26. PMID 23099730
- [Background] Meyer J, Naiken S, Christou N, Liot E, Toso C, Buchs NC, Ris F. Reducing anastomotic leak in colorectal surgery: The old dogmas and the new challenges. World J Gastroenterol. 2019 Sep 14;25(34):5017-5025. doi: 10.3748/wjg.v25.i34.5017. PMID 31558854
- [Background] Carlini M, Grieco M, Spoletini D, Menditto R, Napoleone V, Brachini G, Mingoli A, Marcellinaro R. Implementation of the gut microbiota prevents anastomotic leaks in laparoscopic colorectal surgery for cancer:the results of the MIRACLe study. Updates Surg. 2022 Aug;74(4):1253-1262. doi: 10.1007/s13304-022-01305-6. Epub 2022 Jun 23. PMID 35739383
- [Background] Vasiliu EC, Zarnescu NO, Costea R, Neagu S. Review of Risk Factors for Anastomotic Leakage in Colorectal Surgery. Chirurgia (Bucur). 2015 Jul-Aug;110(4):319-26. PMID 26305194
- [Background] Crafa F, Smolarek S, Missori G, Shalaby M, Quaresima S, Noviello A, Cassini D, Ascenzi P, Franceschilli L, Delrio P, Baldazzi G, Giampiero U, Megevand J, Maria Romano G, Sileri P. Transanal Inspection and Management of Low Colorectal Anastomosis Performed With a New Technique: the TICRANT Study. Surg Innov. 2017 Oct;24(5):483-491. doi: 10.1177/1553350617709182. Epub 2017 May 17. PMID 28514887
- [Background] Ito M, Sugito M, Kobayashi A, Nishizawa Y, Tsunoda Y, Saito N. Relationship between multiple numbers of stapler firings during rectal division and anastomotic leakage after laparoscopic rectal resection. Int J Colorectal Dis. 2008 Jul;23(7):703-7. doi: 10.1007/s00384-008-0470-8. Epub 2008 Apr 1. PMID 18379795
- [Background] Hyman N, Manchester TL, Osler T, Burns B, Cataldo PA. Anastomotic leaks after intestinal anastomosis: it's later than you think. Ann Surg. 2007 Feb;245(2):254-8. doi: 10.1097/01.sla.0000225083.27182.85. PMID 17245179
- [Background] Phitayakorn R, Delaney CP, Reynolds HL, Champagne BJ, Heriot AG, Neary P, Senagore AJ; International Anastomotic Leak Study Group. Standardized algorithms for management of anastomotic leaks and related abdominal and pelvic abscesses after colorectal surgery. World J Surg. 2008 Jun;32(6):1147-56. doi: 10.1007/s00268-008-9468-1. PMID 18283511
- [Background] Alberts JC, Parvaiz A, Moran BJ. Predicting risk and diminishing the consequences of anastomotic dehiscence following rectal resection. Colorectal Dis. 2003 Sep;5(5):478-82. doi: 10.1046/j.1463-1318.2003.00515.x. PMID 12925084
- [Background] Branagan G, Finnis D; Wessex Colorectal Cancer Audit Working Group. Prognosis after anastomotic leakage in colorectal surgery. Dis Colon Rectum. 2005 May;48(5):1021-6. doi: 10.1007/s10350-004-0869-4. PMID 15789125
- [Background] Biondo S, Pares D, Kreisler E, Rague JM, Fraccalvieri D, Ruiz AG, Jaurrieta E. Anastomotic dehiscence after resection and primary anastomosis in left-sided colonic emergencies. Dis Colon Rectum. 2005 Dec;48(12):2272-80. doi: 10.1007/s10350-005-0159-9. PMID 16228841
- [Background] Buchs NC, Gervaz P, Secic M, Bucher P, Mugnier-Konrad B, Morel P. Incidence, consequences, and risk factors for anastomotic dehiscence after colorectal surgery: a prospective monocentric study. Int J Colorectal Dis. 2008 Mar;23(3):265-70. doi: 10.1007/s00384-007-0399-3. Epub 2007 Nov 22. PMID 18034250
- [Background] Platell C, Barwood N, Dorfmann G, Makin G. The incidence of anastomotic leaks in patients undergoing colorectal surgery. Colorectal Dis. 2007 Jan;9(1):71-9. doi: 10.1111/j.1463-1318.2006.01002.x. PMID 17181849
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- [Background] Chadi SA, Fingerhut A, Berho M, DeMeester SR, Fleshman JW, Hyman NH, Margolin DA, Martz JE, McLemore EC, Molena D, Newman MI, Rafferty JF, Safar B, Senagore AJ, Zmora O, Wexner SD. Emerging Trends in the Etiology, Prevention, and Treatment of Gastrointestinal Anastomotic Leakage. J Gastrointest Surg. 2016 Dec;20(12):2035-2051. doi: 10.1007/s11605-016-3255-3. Epub 2016 Sep 16. PMID 27638764
- [Background] van de Velde CJ, Boelens PG, Tanis PJ, Espin E, Mroczkowski P, Naredi P, Pahlman L, Ortiz H, Rutten HJ, Breugom AJ, Smith JJ, Wibe A, Wiggers T, Valentini V. Experts reviews of the multidisciplinary consensus conference colon and rectal cancer 2012: science, opinions and experiences from the experts of surgery. Eur J Surg Oncol. 2014 Apr;40(4):454-68. doi: 10.1016/j.ejso.2013.10.013. Epub 2013 Nov 8. PMID 24268926
- [Background] van de Velde CJ, Boelens PG, Borras JM, Coebergh JW, Cervantes A, Blomqvist L, Beets-Tan RG, van den Broek CB, Brown G, Van Cutsem E, Espin E, Haustermans K, Glimelius B, Iversen LH, van Krieken JH, Marijnen CA, Henning G, Gore-Booth J, Meldolesi E, Mroczkowski P, Nagtegaal I, Naredi P, Ortiz H, Pahlman L, Quirke P, Rodel C, Roth A, Rutten H, Schmoll HJ, Smith JJ, Tanis PJ, Taylor C, Wibe A, Wiggers T, Gambacorta MA, Aristei C, Valentini V. EURECCA colorectal: multidisciplinary management: European consensus conference colon & rectum. Eur J Cancer. 2014 Jan;50(1):1.e1-1.e34. doi: 10.1016/j.ejca.2013.06.048. Epub 2013 Oct 31. PMID 24183379
- [Background] Hermanek P Jr, Wiebelt H, Riedl S, Staimmer D, Hermanek P. [Long-term results of surgical therapy of colon cancer. Results of the Colorectal Cancer Study Group]. Chirurg. 1994 Apr;65(4):287-97. German. PMID 8020349
- [Background] Ferlay J, Ervik M, Lam F, Laversanne M, Colombet M, Mery L, et al. https://gco.iarc.who.int/today. 2024. Global Cancer Observatory: Cancer Today (version 1.1). Lyon, France: International Agency for Research on Cancer. Available from: https://gco.iarc.who.int/today
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT07099820/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT07099820/ICF_001.pdf